CLINICAL TRIAL: NCT03765372
Title: Evaluation of hsTnT for Perioperative Risk Stratification Among Patients Undergoing Elective Non-cardiac Surgery
Brief Title: Evaluation of BIomarkers for POstoperative Complications in Non-cardiac Surgery Patients
Status: Completed | Type: Observational
Sponsor: Technical University of Munich (Other)
Responsible Party: Sponsor
Other Study IDs: BiPoC
Record Dates: First submitted 2018-11-28; First posted 2018-12-05 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2021-12

CONDITIONS: Perioperative/Postoperative Complications; Outcome
Keywords: perioperative outcome; clavien-dindo classification; hsTnT; MINS
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Weeks
Biospecimen Retention: Samples Without DNA — blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Aim of this study is to evaluate whether the periopertive course is able to predict postoperative complications. Several approaches will be choosed to optimize perioperative risk stratification predicting postoperative complications in patients undergoing elective non-cardiac surgery.

DETAILED DESCRIPTION:
The aim of this secondary analysis of the SUPERADD study is to use the perioperative data from the prospective SUPERADD study ("SUbstitution of PERioperative Albumin Deficiency Disorders") (Eudra-CT 2016-001313-24; Clinical Trials NCT03167645; DOI: 10.1097) to identify risk factors for the occurrence of postoperative complications, based on the Clavien-Dindo classification in the nine domains of the Postoperative Morbidity Survey.

Multivariate Analyses, Decision trees, time series analysis and Machine Learning methods will be applied to distinguish risk factors for postoperative complikations and mortality in a high-risk group (see publication of the statistical analysis plan and its enhancement).

Patients participating in the SUPERADD study (NCT03167656) and who had at least two perioperative high sensitive Troponin T (hsTnT) values in order to detect myocardial injury were included in this secondary analysis as hsTnT is associated with major adverse cardiovascular events (MACE), myocardial injury after noncardiac surgery and mortality.

The secondary analysis uses data obtained at the pre-anaesthesia visit like ASA, preoperative comorbidities measured by the POSPOM, CCI, intraoperative parameters like vitals, medication, estimated blood loss and postoperative data obtained from PACU records and discharge letter. Primary Endpoint are postoperative complications assessed with the Cavien-Dindo classification > 2.

ELIGIBILITY:
Inclusion Criteria:

* written informed consense
* Age > 18 years
* ASA Score 3 or 4
* elective non-cardiac high risk surgery

Exclusion Criteria:

* emergency surgery
* need for dialysis
* liver cirrhosis child C
* intolerance of albumin
* participation in other AMG (medicines law) study
* pregnancy or breastfeeding
* patients with attendants concerning medical matters
* ASA V patients
* patients with BMI > 35 kg/m2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: High risk patients (ASA Status 3 or 4) and / or patients undergoing elective non-cardiac high risk surgery at the Klinikum rechts der Isar, Munich.
Sampling Method: Probability Sample
Enrollment: 1598 (Actual)
Dates: Start 2017-06-19 (Actual); Primary Completion 2019-11-01 (Actual); Study Completion 2021-12-18 (Actual)

PRIMARY OUTCOMES:
postoperative complications determined with the calvien-dindo classification | date of surgery until hospital discharge (approx. 30 days)
  Pulmonary, infectious, renal, gastrointestinal, cardiovascular, neurological, wound, haematological and pain. Each domain is graded between grade I and V (death of a patient).

SECONDARY OUTCOMES:
hospital mortality | date of surgery until hospital discharge (approx. 30 days)
  Rate of Mortality among study patients
Acute Kidney Injury | postoperative day 2
  Acute Kidney Injury according to KDIGO
Myocardial Injury | postoperative day 2
  perioperative hsTnT course, including preoperative hsTnT measurements
6 months mortalitiy | date of surgery until 6 months after
  Rate of Mortality among study patients

CONTACTS AND LOCATIONS:
Overall Officials: Bettina Jungwirth, Prof., Study Director — Department of Anesthesia, Klinikum rechts der Isar, TU Munich
Locations (1):
- Klinikum Rechts der Isar, Technische Universität München, München, Bavaria, Germany

REFERENCES:
- [Result] Anetsberger A, Blobner M, Haller B, Schmid S, Umgelter K, Hager T, Langgartner C, Kochs EF, Laugwitz KL, Jungwirth B, Bernlochner I. Immature platelets as a novel biomarker for adverse cardiovascular events in patients after non-cardiac surgery. Thromb Haemost. 2017 Oct 5;117(10):1887-1895. doi: 10.1160/TH16-10-0804. Epub 2017 Aug 10. PMID 28796275
- [Result] Writing Committee for the VISION Study Investigators; Devereaux PJ, Biccard BM, Sigamani A, Xavier D, Chan MTV, Srinathan SK, Walsh M, Abraham V, Pearse R, Wang CY, Sessler DI, Kurz A, Szczeklik W, Berwanger O, Villar JC, Malaga G, Garg AX, Chow CK, Ackland G, Patel A, Borges FK, Belley-Cote EP, Duceppe E, Spence J, Tandon V, Williams C, Sapsford RJ, Polanczyk CA, Tiboni M, Alonso-Coello P, Faruqui A, Heels-Ansdell D, Lamy A, Whitlock R, LeManach Y, Roshanov PS, McGillion M, Kavsak P, McQueen MJ, Thabane L, Rodseth RN, Buse GAL, Bhandari M, Garutti I, Jacka MJ, Schunemann HJ, Cortes OL, Coriat P, Dvirnik N, Botto F, Pettit S, Jaffe AS, Guyatt GH. Association of Postoperative High-Sensitivity Troponin Levels With Myocardial Injury and 30-Day Mortality Among Patients Undergoing Noncardiac Surgery. JAMA. 2017 Apr 25;317(16):1642-1651. doi: 10.1001/jama.2017.4360. PMID 28444280
- [Result] Ma J, Xin Q, Wang X, Gao M, Wang Y, Liu J. Prediction of perioperative cardiac events through preoperative NT-pro-BNP and cTnI after emergent non-cardiac surgery in elderly patients. PLoS One. 2015 Mar 23;10(3):e0121306. doi: 10.1371/journal.pone.0121306. eCollection 2015. PMID 25799524
- [Result] Vetrugno L, Costa MG, Pompei L, Chiarandini P, Drigo D, Bassi F, Gonano N, Muzzi R, Della Rocca G. Prognostic power of pre- and postoperative B-type natriuretic peptide levels in patients undergoing abdominal aortic surgery. J Cardiothorac Vasc Anesth. 2012 Aug;26(4):637-42. doi: 10.1053/j.jvca.2012.01.018. Epub 2012 Mar 2. PMID 22387082